CLINICAL TRIAL: NCT02665663
Title: Measure of the Strength of the Tongue in Patients With Amyotrophic Lateral Sclerosis and Relation With Swallowing Disorders
Brief Title: Tongue Strength in Amyotrophic Lateral Sclerosis (ALS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2015-18
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- healthy volunteers (Other): Constitution of a control group consisting of 20 healthy volunteers, matched for age and sex to establish a "normal" pressure force of the language depending on the age and sex value
  Interventions: Device: medical device
- Patients with Amyotrophic Lateral Sclerosis (Other): Constitution of a group of 20 patients with Amyotrophic Lateral Sclerosis (ALS), included at diagnosis of the disease on clinical and electromyographic arguments addressed in speech pathology consultation without a complaint swallowing.
  Interventions: Device: medical device
- patients with Amyotrophic Lateral Sclerosis and swallowi (Other): Constitution of a group of 20 patients with Amyotrophic Lateral Sclerosis ( ALS) and swallowing disorders clinically objectified in the ENT consultation.
  Interventions: Device: medical device

INTERVENTIONS:
Device: medical device

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is a neurodegenerative disease with a poor prognosis that occurs in adults 64 years on average. Its prevalence is 4 to 6/100 000 inhabitants.

Swallowing disorders occur during evolution and involve the prognosis of patients in the short term by the association of dysphagia with severe malnutrition, and aspiration. The issue of phoniatric monitoring is to detect early onset of the swallowing disorders to develop strategies for respiratory protection, food adapted to disturbances, and speech therapy.

The objective of this study is to compare the tongue force in patients with amyotrophic lateral sclerosis at the time of diagnosis and at the onset of swallowing disorders compared to healthy subjects, with the dynamic palatography device developed in the Laboratoire Parole et Langage (UMR 7309, CNRS-Université Aix-Marseille, Aix-en-Provence), which allows the measurement of the strength and duration of the pression of the tongue on the palate.

ELIGIBILITY:
Inclusion Criteria:

* Adults and legally responsible/ valid medical insurance
* patients : ALS diagnostic already announced
* healthy subjects : EAT-10 score<2

Exclusion Criteria:

* Non pregnant and non baby feeding
* Presence of risk factor or suspicion of Creutzfeld Jacob Disease
* Allergy/intolerance to the glueing paste
* Antecedent of pathology of the aerodigestive tract
* Other neurologic disease
* Morphologic anomaly of the aerodigestive tract
* Excessive gag reflex

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-03 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Maximum tongue strength | 30 minutes
  maximal tongue strength during salivary swallowing
Tongue contact duration | 30 minutes
  Duration of tongue and palate contact during salivary

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Service ORL Assistance Publique Hôpitaux de Marseille, Marseille, France